CLINICAL TRIAL: NCT03248765
Title: Human Brain Adaptation to Chronic Pain and Its Effects on Opioid Use
Status: Terminated | Type: Observational
Why Stopped: Insufficient patient enrollment.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201707017
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Pain, Chronic; Opioid Use
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genotype analysis will be performed to control for A118G single nucleotide polymorphism (SNP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic pain group: post-surgical opioid use measured at 1 day and 1 week.
  Interventions: Other: post-surgical opioid use measured at 1 day and 1 week.
- No chronic pain: post-surgical opioid use measured at 1 day and 1 week.
  Interventions: Other: post-surgical opioid use measured at 1 day and 1 week.

INTERVENTIONS:
Other: post-surgical opioid use measured at 1 day and 1 week. — Evaluation of intra-hospital perioperative opioid administration (including intraoperative opioids and Patient Controlled Analgesia (PCA) use). This endpoint is calculated as the total amount of morphine equivalents administered intraoperatively and in the first 24 hours after the end surgery (measured on postoperative day 1).
  2) Opioid utilization after discharge from hospital (prescription refills and pills count at subsequent hospital visits). This endpoint is calculated as the total amount of morphine equivalents consumed in the first week after the surgery (measured at 1 week after surgery by electronic questionnaire and verified by direct pill count performed on occasion of the patient's postsurgical visit ).

SUMMARY:
The purpose of this study is to determine if the research results obtained in animal models of pain - that show that being in pain for some time increases opioid use beyond what is expected to treat the current pain - also apply to patients with chronic pain.

DETAILED DESCRIPTION:
The prevalence of chronic pain is very high in the US at approximately 30%. More than 10% of adults report having daily pain. Opioid pain medications [such as morphine] are prescribed for some pain conditions and, since they are very addictive, they can be used inappropriately and abused, to the point of causing overdose and death. This is currently a significant problem in the US and worldwide. Research on changes in the brain that cause addiction in pain patients is complicated, also because it is difficult to separate the effect of the drugs that cause addiction from the direct effect of pain on the brain. Studies in animals have found that pain per se can change the brain in ways that increase the risk of becoming addicted to pain medications. Therefore, we think that patients who have chronic pain and are prescribed opioid pain medications to treat surgery-related pain after surgery, although they never took opioids for a long time in their life, may be at increased risk of using too much opioid medications, and using opioids for a longer time than expected to treat their surgical pain.

The purpose of this study is to determine if the research results obtained in animal models of pain (that show that being in pain for some time increases opioid use beyond what is expected to treat the current pain) also apply to patients with chronic pain.

For our study we are looking to recruit patients scheduled for abdominal surgery at Barnes Jewish Hospital. If eligible and enrolled, subjects will undergo sensory testing (a test of the sensitivity of the skin to hot and cold temperature and pressure) and complete questionnaires about their experience with pain, anxiety, depression and risk of substance abuse. They will also have a one-time blood draw for genetic testing, to look for a particular gene that is potentially associated with how we respond to pain medications and, potentially, with increased risk for addiction. After the surgery, patients will be assessed by the research team on day 1, week 1, week 4, week 8, and after 6 months with similar questionnaires to those that were completed pre-surgery. Patient satisfaction with their pre-surgical and post-surgical pain control will also be assessed by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. With and without history of chronic muscle-skeletal pain *
3. Scheduled to undergo elective abdominal surgery requiring overnight hospital admission
4. Opioid naïve**
5. Willing to comply with study procedures as outlined in the protocol
6. Willing and able to provide informed consent
7. Having an email address and access to a computer or electronic tablet

Exclusion Criteria:

1. Current use of opioids (includes ANY use in past 3 months)
2. Cancer diagnosis
3. Patient presenting the following documented conditions:

Untreated psychosis Current suicidal ideation Current substance abuse

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with and without chronic musculoskeletal pain or osteoarthritis pain that are having planned non-cancer related surgery
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Post-surgical opioid use | 24 hours post-operatively
  oral morphine equivalents (mg/day)
Post-surgical opioid use | 1 week post-operatively
  oral morphine equivalents (mg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Cavallone, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided